CLINICAL TRIAL: NCT02861599
Title: Study of the Interest of Proprioceptive Therapy as a Complement to Speech Therapy in Children With Reading Difficulties
Acronym: 2000DYS9
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: QUERCIA INSERM 2015
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-07

CONDITIONS: Reading Difficulties
MeSH Terms: interventions — Speech Therapy

ARMS (2):
- proprioceptive therapy (Experimental)
  Interventions: Other: proprioceptive therapy; Other: speech therapy
- speech therapy (Placebo Comparator)
  Interventions: Other: speech therapy

INTERVENTIONS:
Other: proprioceptive therapy
  Arms: proprioceptive therapy
Other: speech therapy

SUMMARY:
Before proposing this observational study protocol, a randomized study was attempted. This consisted in proposing to families of children with difficulties in learning to read, via the speech therapists who were treating them, to take part in a randomized trial that compared speech therapy alone with a combination of speech therapy and proprioceptive therapy. If parents agreed in principle with the study, the child underwent a complementary speech therapy examination and was referred to the nearest investigating doctor for inclusion. However, this study had to be abandoned because of insufficient recruitment (2 patients included in 1 year). Despite the motivation and training of participating speech therapists, proposing a study based on randomization to families often in distress proved to be extremely difficult, as their conviction of the interest of proprioceptive therapy was greater than the available scientific evidence suggested. Direct recruitment by investigating ophthalmologists was not possible because they were consulted directly by the families so as to obtain proprioceptive therapy. The principle of randomization would thus not have been accepted.

In light of the above, we decided to turn towards a non-randomized study comparing outcomes in two groups of children:

* children who consulted an ophthalmologist who proposed proprioceptive therapy in Côte d'Or
* children managed by one of the four speech therapists who do not propose proprioceptive therapy and who accepted the principle of the study.

ELIGIBILITY:
Inclusion Criteria:

For both groups:

* children at school and between the end of year 3 and the end of year 7
* with speech therapy for reading difficulties
* with a delay of 18 months or more compared with children in the same group at inclusion
* who had never had proprioceptive therapy
* in cases of two or more siblings with reading difficulties between year 3 and year 8, only one child will be included.
* With one speech therapy session per week
* Who have accepted to take part in the study in agreement with their parents
* With national health insurance cover For the " speech therapy only" cohort: children followed by speech therapists who do not usually refer their patients to ophthalmologists that use proprioceptive therapy in cases of delayed reading acquisition and have not previously consulted an ophthalmologist proposing this type of therapy.

For the " speech therapy associated with proprioceptive therapy " cohort: children with reading difficulties followed by a speech therapist and consulting for the first time an ophthalmologist, study investigator, who uses proprioceptive therapy in the treatment of reading difficulties.

Exclusion Criteria:

* Children who lack motivation and/or and those unlikely to be followed in optimal conditions
* Neonatal distress: APGAR <7
* Gestational age < 37 weeks of Amenorrhea (WA)
* Genetic disease
* Known abnormal or delay in psychomotor development
* Psychiatric disorder
* Sensory deficit or disorder known to limit the possibilities of proprioceptive therapy
* Children undergoing treatment, notably psychotropic agents, Ritaline®, antiepileptic agents or rehabilitation, which may interfere with reading difficulties or the therapy proposed in the study
* Children in special needs schools (SEGPA)
* Children who cannot attend all of the consultations planned in the protocol for practical reasons.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of children who had stabilized their delay in reading acquisition at the Timé-3 test (identification of written words) | At month12

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France